CLINICAL TRIAL: NCT03250325
Title: Multi-center Phase I/II Study of NY-ESO-1 T Cell Receptor Gene Transferred T Lymphocytes in Patients with Synovial Sarcoma
Brief Title: Study of TBI-1301 (NY-ESO-1 T Cell Receptor Gene Transduced Autologous T Lymphocytes) in Patients with Synovial Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1301-03
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Synovial Sarcoma
Keywords: Adoptive cell transfer; Cell therapy; Immunotherapy; NY-ESO-1; T cell receptor gene therapy; Synovial sarcoma
MeSH Terms: conditions — Sarcoma, Synovial | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Split dose of 5x10^9 TBI-1301 (Experimental): Split dose of 5x10^9 TBI-1301 will be administered intravenously for 2 days following cyclophosphamide pre-treatment 750 mg/m2/d for 2 days.
  Interventions: Biological: TBI-1301; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TBI-1301 — Split dose of TBI-1301 is administered intravenously for 2 days following cyclophosphamide pre-treatment.
Drug: Cyclophosphamide — Cyclophosphamide (750mg/m2/day x 2 days Intravenous (IV)) is administered as pre-treatment medication of TBI-1301.

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of TBI-1301 for NY-ESO-1 expressing synovial sarcoma when administered following cyclophosphamide pre-treatment.

DETAILED DESCRIPTION:
Following pre-treatment with cyclophosphamide, NY-ESO-1-specific T cell receptor (TCR) gene transduced T lymphocytes are transferred to human leukocyte antigen (HLA)-A*02:01 or HLA-A*02:06 positive patients with synovial sarcoma expressing NY-ESO-1, which are surgically unresectable and refractory to anthracycline therapy. The primary objective is to evaluate the safety in the phase 1 and the efficacy in the phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed synovial sarcoma
2. Surgically unresectable tumor
3. Progressing or recurrent synovial sarcoma which has been treated with 1-4 regimens of systemic chemotherapies including anthracycline
4. HLA-A*02:01 or HLA-A*02:06 positive
5. Tumor that express NY-ESO-1 by immunohistochemistry
6. ≥ 18 years of age
7. Measurable lesions that are evaluable by the RECIST ver1.1
8. ECOG Performance Status of 0, 1 or 2
9. No treatment such as chemotherapy and be expected to recover fully from the previous treatment at the time of the lymphocytes collection for manufacturing
10. Life expectancy ≥ 16 weeks after consent
11. No severe damage on the major organs (bone marrow, heart, lung, liver, kidney, etc) and meet the following lab value criteria; Total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST(GOT), ALT(GPT) < 3.0 x ULN; Creatinine < 1.5 x ULN; 2,500/μL < WBC ≤ULN; Hemoglobin ≥ 8.0g/dL; Platelets ≥ 75,000/μL
12. Patients must be able to understand the study contents and to give a written consent at his/her free will. Additionally, if patients are below 20 years of age, proxies must be able to give a written consent.

Exclusion Criteria:

1. Patients with the following conditions are excluded from the study; Unstable angina, cardiac infarction, or heart failure; Uncontrolled diabetes or hypertension; Active infection; Obvious interstitial pneumonia or lung fibrosis by chest X-ray; Active autoimmune disease requiring steroids or immunosuppressive therapy.
2. Active metastatic tumor cell invasion into CNS
3. Active multiple cancer
4. Positive for HBs antigen or HBV-DNA observed in serum
5. Positive for HCV antibody and HCV-RNA observed in serum
6. Positive for antibodies against HIV or HTLV-1
7. Left Ventricular Ejection Fraction (LVEF) ≤ 50%
8. History of serious hypersensitivity reactions to bovine or murine derived substances.
9. History of hypersensitivity reaction to ingredients or excipients of investigational drugs used in this study
10. History of hypersensitivity reaction to antibiotics used in manufacturing for the investigational drug used in this study.
11. Pregnant females, lactating females (except when they cease and do not resume lactation) or female and male patients who cannot agree to practice the adequate birth control from the consent to 6 months after infusion of the investigational drug.
12. Clinically significant systemic illness that in the judgment of the PI or sub-investigator would compromise the patient's ability to tolerate protocol therapy or significantly increase the risk of complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
(Phase I) Adverse event, mortality, severe adverse event, discontinuation due to adverse event, laboratory test values | 52 weeks
  Confirm the toxicity profile, which is measured by the degree of grade and seriousness, duration, causality, classification, etc. of the adverse events.
(Phase I) Appearance of replication competent retrovirus (RCR) by PCR | 52 weeks
  Confirm that no replication competent retrovirus observed.
(Phase I) Appearance of clonality by linear amplification mediated (LAM)-PCR | 52 weeks
  Confirm that no clonality is observed.
(Phase I) Blood kinetics of TBI-1301 by realtime-PCR | 52 weeks
  Evaluate persistence and expansion of transferred TBI-1301.
(Phase II) Overall response rate | 52 weeks
  Evaluate response rate by measuring response using RECIST v1.1 and irRECIST

SECONDARY OUTCOMES:
(Phase I) Objective response rate | 52 weeks
  Evaluate response rate by measuring response using RECIST v1.1 and irRECIST
(Phase I/II) Progression free rate | 12 weeks
  Evaluate progression free rate by measuring response using RECIST v1.1 and irRECIST
(Phase I/II) Progression free survival | 52 weeks
  Evaluate progression free survival
(Phase I/II) Overall survival | 52 weeks
  Evaluate overall survival
(Phase II) Adverse event, mortality, severe adverse event, discontinuation due to adverse event, laboratory test values | 52 weeks
  Confirm the toxicity profile, which is measured by the degree of grade and seriousness, duration, causality, classification, etc. of the adverse events.
(Phase II) Appearance of RCR | 52 weeks
  Confirm that no replication competent retrovirus observed.
(Phase II) Appearance of clonality (LAM-PCR) | 52 weeks
  Confirm that no clonality is observed.
(Phase II) Blood kinetics of TBI-1301 by realtime-PCR | 52 weeks
  Evaluate persistence and expansion of transferred TBI-1301.

CONTACTS AND LOCATIONS:
Overall Officials: Masanobu Kimura, Study Director — Takara Bio Inc.
Locations (5):
- Japan (5):
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Mie University Hospital, Tsu, Mie-ken
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: Undecided